CLINICAL TRIAL: NCT06550154
Title: Association Between Oral Lichen Planus and Thyroid Disease: A Cross-sectional Study
Brief Title: Association Between Oral Lichen Planus and Thyroid Disease
Status: Completed | Type: Observational
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Stephanie Rodríguez-Fernández, Principal Investigator, University of Barcelona
Other Study IDs: 2024-001-1
Record Dates: First submitted 2024-08-05; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Oral Lichen Planus; Thyroid Disease
Keywords: oral lichen planus; thyroid disease; thyroid disorders; hypothyroidism; arterial hypertension; dyslipidemia; diabetes mellitus; depression; anxiety; association; prevalence
MeSH Terms: conditions — Lichen Planus, Oral; Thyroid Diseases; Hypothyroidism; Hypertension; Dyslipidemias; Diabetes Mellitus; Depression; Anxiety Disorders | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- OLP patients: 60 subjects with oral lichen planus
  Interventions: Other: Data collection
- Control group: 60 subjects without oral lichen planus. Each control subject was matched by age and sex to its corresponding paired OLP subject
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Participants were identified by reviewing electronic medical records. Medical history information of thyroid disease and associated medication were collected in both groups, as well as a history of other comorbidities such as diabetes mellitus type 2, arterial hypertension, dyslipidemia, anxiety, and depression. Cases and controls were matched by age and sex.

SUMMARY:
The goal of this observational study is to determine the prevalence of thyroid disease in adults with oral lichen planus (OLP) treated at the Dental Hospital of the University of Barcelona (HOUB), and to evaluate the association between OLP and thyroid disease. Secondly, to assess the association between OLP and other comorbidities, including arterial hypertension, diabetes mellitus type 2, dyslipidemia, anxiety, and depression.

The main question it aims to answer is: Do people with OLP have a significant risk of developing thyroid disorders compared to people without OLP?

DETAILED DESCRIPTION:
A cross-sectional study was conducted to investigate a total of 120 participants, 60 patients with oral lichen planus and 60 patients without the history of OLP as a control group, attending at the Dental Hospital of the University of Barcelona (HOUB). The personal medical history of thyroid disease, demographic information (age and gender) and other comorbidities history information, were collected in both groups, and obtained through the GESDEN® healthcare software (Gesden G5, Infomed - Henry Schein®, New York, United States), in addition to the paper medical records (biopsy report). Data were analyzed using χ² test and simple binary logistic regression models with the SPSS® statistical software, version 29.0.2.0 for Windows (SPSS, Illinois, United States).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* For the case group: patients with OLP clinically and histologically diagnosed according to the diagnostic criteria of the American Academy of Oral and Maxillofacial Pathology.
* For the control group: patients without OLP lesions, who came to the HOUB for the treatment of other oral pathologies, and who also do not have a history of clinically and histologically diagnosed OLP.

Exclusion Criteria:

* Patients under 18 years of age.
* Patients with lichenoid lesions induced by drug reactions or by contact with restorative materials such as amalgam.
* Patients with complicated or uncontrolled systemic diseases.
* Patients with other autoimmune diseases (such as systemic lupus erythematosus, Sjögren's syndrome, rheumatoid arthritis, psoriasis, celiac disease, vitiligo, diabetes mellitus type 1).
* Pregnant patients.

Ages: 29 Years to 94 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients who attended the Dental Hospital of the University of Barcelona (HOUB).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Prevalence of thyroid disease in patients with OLP | 1 day
  Percentage of patients with OLP who have thyroid disease, determined through the review of medical records. Prevalence refers to the number of existing cases at the time of the study, reflecting the proportion of individuals with thyroid disease among the patients evaluated. Outcomes are presented in frequencies and percentages. The χ² test was used to compare the categorical variables. All the analysis was carried out on SPSS.
Prevalence of the most common thyroid disorders | 1 day
  Determine which thyroid disorder is most common in the study population. Outcomes are presented in frequencies and percentages. All the analysis was carried out on SPSS.
Association between OLP and thyroid disease | 1 day
  It is determined by comparing the frequency of thyroid disease in patients with OLP versus controls, using statistical analysis (binary logistic regression) to assess the strength and significance of such association. All the analysis was carried out on SPSS.

SECONDARY OUTCOMES:
Distribution of OLP according age and gender | 1 day
  Frequency and percentage of OLP in different age ranges and both sexes to identify potential prevalence patterns associated with these demographic factors. Outcomes are presented in frequencies, percentages and mean ± standard deviation. All the analysis was carried out on SPSS.
Prevalence of other comorbidities analyzed (arterial hypertension, diabetes mellitus type 2, dyslipidemia, anxiety, and depression) | 1 day
  Prevalence reflects the proportion of individuals affected by each pathology at the time of evaluation. Outcomes are presented in frequencies and percentages. The χ² test was used to compare the categorical variables. All the analysis was carried out on SPSS.
Association between OLP and other comorbidities analyzed (arterial hypertension, diabetes mellitus type 2, dyslipidemia, anxiety, and depression) | 1 day
  This involves determining whether there is a significant association between OLP and these comorbidities in the study population. Statistical analysis (binary logistic regression) evaluates the strength and significance of such associations to identify potential risk factors related to OLP. All the analysis was carried out on SPSS.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Rodríguez-Fernández, Principal Investigator — University of Barcelona; Sonia Egido-Moreno, Principal Investigator — University of Barcelona; José López López, Principal Investigator — University of Barcelona
Locations (1):
- Campus Bellvitge, Facultat de Medicina i Ciències de la Salut, Universitat de Barcelona, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data. Data are available indefinitely. Proposals should be directed to stephroferd@gmail.com

REFERENCES:
- [Background] Maddheshiya N, Shivakumar GC, Misra N, Rastogi V, Kumar S. Prevalence of oral lichen planus in patients with hypothyroidism versus non-hypothyroidism - A case control study of 1000 cases. J Oral Maxillofac Pathol. 2022 Oct-Dec;26(4):509-517. doi: 10.4103/jomfp.jomfp_517_20. Epub 2022 Dec 22. PMID 37082069
- [Background] Zhang T, Hou F, Liu D, Zhou H, Sun Y, Deng X, Xu Y, Xiao Y, Wang X, Wu C, Meng Y, Yuan P, Qiu X, Ye L, Liang Y, Wei W, Jiang L. Association of Hashimoto's thyroiditis and anti-thyroid antibodies with oral lichen planus: A cross-sectional study. Front Immunol. 2022 Aug 16;13:967988. doi: 10.3389/fimmu.2022.967988. eCollection 2022. PMID 36052085
- [Background] Wang Y, Hao Y, Tang F, Chen Q. Immune mechanisms involved in the coexistence of oral lichen planus and autoimmune thyroid diseases. Zhejiang Da Xue Xue Bao Yi Xue Ban. 2021 Apr 25;50(2):222-228. doi: 10.3724/zdxbyxb-2021-0124. PMID 34137220
- [Background] Shahid MA, Ashraf MA, Sharma S. Physiology, Thyroid Hormone. 2023 Jun 5. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK500006/ PMID 29763182
- [Background] Siponen M, Huuskonen L, Laara E, Salo T. Association of oral lichen planus with thyroid disease in a Finnish population: a retrospective case-control study. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Sep;110(3):319-24. doi: 10.1016/j.tripleo.2010.04.001. Epub 2010 Jul 24. PMID 20656530
- [Background] Alikhani M, Ghalaiani P, Askariyan E, Khunsaraki ZA, Tavangar A, Naderi A. Association between the clinical severity of oral lichen planus and anti-TPO level in thyroid patients. Braz Oral Res. 2017 Jan 5;31:e10. doi: 10.1590/1807-3107BOR-2017.vol31.0010. PMID 28076499
- [Background] Li D, Li J, Li C, Chen Q, Hua H. The Association of Thyroid Disease and Oral Lichen Planus: A Literature Review and Meta-analysis. Front Endocrinol (Lausanne). 2017 Nov 9;8:310. doi: 10.3389/fendo.2017.00310. eCollection 2017. PMID 29170653
- [Background] De Porras-Carrique T, Ramos-Garcia P, Aguilar-Diosdado M, Warnakulasuriya S, Gonzalez-Moles MA. Autoimmune disorders in oral lichen planus: A systematic review and meta-analysis. Oral Dis. 2023 May;29(4):1382-1394. doi: 10.1111/odi.14127. Epub 2022 Feb 1. PMID 35000260
- [Background] Garcia-Pola MJ, Llorente-Pendas S, Seoane-Romero JM, Berasaluce MJ, Garcia-Martin JM. Thyroid Disease and Oral Lichen Planus as Comorbidity: A Prospective Case-Control Study. Dermatology. 2016;232(2):214-9. doi: 10.1159/000442438. Epub 2016 Jan 20. PMID 26784745
- [Background] Robledo-Sierra J, Landin-Wilhelmsen K, Filipsson Nystrom H, Eggertsen R, Larsson L, Dafar A, Warfvinge G, Mattsson U, Jontell M. A mechanistic linkage between oral lichen planus and autoimmune thyroid disease. Oral Dis. 2018 Sep;24(6):1001-1011. doi: 10.1111/odi.12850. Epub 2018 May 29. PMID 29500871
- [Background] Arduino PG, Karimi D, Tirone F, Sciannameo V, Ricceri F, Cabras M, Gambino A, Conrotto D, Salzano S, Carbone M, Broccoletti R. Evidence of earlier thyroid dysfunction in newly diagnosed oral lichen planus patients: a hint for endocrinologists. Endocr Connect. 2017 Nov;6(8):726-730. doi: 10.1530/EC-17-0262. PMID 29101247
- [Background] Wu P, Luo S, Zhou T, Wang R, Qiu X, Yuan P, Yang Y, Han Q, Jiang L. Possible Mechanisms Involved in the Cooccurrence of Oral Lichen Planus and Hashimoto's Thyroiditis. Mediators Inflamm. 2020 Feb 4;2020:6309238. doi: 10.1155/2020/6309238. eCollection 2020. PMID 32089646
- [Background] Piloni S, Ferragina F, Barca I, Kallaverja E, Cristofaro MG. The Correlation between Oral Lichen Planus and Thyroid Pathologies: A Retrospective Study in a Sample of Italian Population. Eur J Dent. 2024 May;18(2):510-516. doi: 10.1055/s-0043-1772247. Epub 2023 Sep 20. PMID 37729935
- [Background] Cheng YS, Gould A, Kurago Z, Fantasia J, Muller S. Diagnosis of oral lichen planus: a position paper of the American Academy of Oral and Maxillofacial Pathology. Oral Surg Oral Med Oral Pathol Oral Radiol. 2016 Sep;122(3):332-54. doi: 10.1016/j.oooo.2016.05.004. Epub 2016 Jul 9. PMID 27401683
- [Background] Zhou T, Li D, Chen Q, Hua H, Li C. Correlation Between Oral Lichen Planus and Thyroid Disease in China: A Case-Control Study. Front Endocrinol (Lausanne). 2018 Jun 18;9:330. doi: 10.3389/fendo.2018.00330. eCollection 2018. PMID 29967591
- [Background] Kats L, Goldman Y, Kahn A, Goldman V, Gorsky M. Oral lichen planus and thyroid gland diseases: possible associations. BMC Oral Health. 2019 Jul 31;19(1):169. doi: 10.1186/s12903-019-0859-5. PMID 31366342
- [Background] Hasan S, Ahmed S, Kiran R, Panigrahi R, Thachil JM, Saeed S. Oral lichen planus and associated comorbidities: An approach to holistic health. J Family Med Prim Care. 2019 Nov 15;8(11):3504-3517. doi: 10.4103/jfmpc.jfmpc_749_19. eCollection 2019 Nov. PMID 31803644
- [Background] De Porras-Carrique T, Ramos-Garcia P, Gonzalez-Moles MA. Hypertension in oral lichen planus: A systematic review and meta-analysis. Oral Dis. 2024 May;30(4):1793-1805. doi: 10.1111/odi.14727. Epub 2023 Sep 19. PMID 37725328
- [Background] Dave A, Shariff J, Philipone E. Association between oral lichen planus and systemic conditions and medications: Case-control study. Oral Dis. 2021 Apr;27(3):515-524. doi: 10.1111/odi.13572. Epub 2020 Aug 20. PMID 32750751
- [Background] Li KY, Li CL, Hua H, Song ZF. Potential relationship of dyslipidemia with dietary patterns in oral lichen planus patients-A case-control study. J Dent Sci. 2023 Oct;18(4):1638-1644. doi: 10.1016/j.jds.2023.01.006. Epub 2023 Feb 11. PMID 37799923
- [Background] Vallejo MJ, Huerta G, Cerero R, Seoane JM. Anxiety and depression as risk factors for oral lichen planus. Dermatology. 2001;203(4):303-7. doi: 10.1159/000051777. PMID 11752817